CLINICAL TRIAL: NCT00998543
Title: A Long-Term Safety and Immunogenicity Follow-up of Healthy Adults Vaccinated With One Dose of Smallpox Vaccine (LISTER Strain)
Brief Title: A Long-Term Study of Healthy Adults Vaccinated With One Dose of Smallpox Vaccine (LISTER Strain)
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: VVL05
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Smallpox
Keywords: Smallpox Vaccinia Virus Smallpox Vaccine Variola Virus
MeSH Terms: conditions — Smallpox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Smallpox Vaccine (LISTER Strain) Group: Participants were vaccinated with the second-generation smallpox vaccine in Study VVL04 (NCT 00258947).

SUMMARY:
The purpose of this study is to provide long-term follow-up immunogenicity and safety data on participants who were vaccinated with the second-generation smallpox vaccine in Study VVL04 (NCT 00258947).

Primary Objectives:

Immunogenicity: To yearly describe the vaccinia antibody persistence up to 5 years post-vaccination.

Safety: To follow-up the long-term safety up to 5 years post-vaccination.

DETAILED DESCRIPTION:
None of the participants in this study will receive any vaccination as part of the study. All participants will provide blood samples for immunogenicity testing at the 1, 2, 3, 4, and 5 year anniversaries of vaccination. Safety will be assessed for up to 5 years after vaccination, including follow-up of reactions that occurred during Study VVL04 (NCT 00258947).

ELIGIBILITY:
Inclusion Criteria :

* Subject vaccinated and who completed the Phase II VVL04 trial.
* Informed consent form signed.
* Subject able to comply with all trial procedures.
* Subject entitled to national social security.

Exclusion Criteria :

* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants were vaccinated with the second-generation smallpox vaccine in Study VVL04 (NCT 00258947)
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2006-10; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immune response of live vaccinia virus (LISTER strain) after primary vaccination. | 1 to 5 years post-vaccination
To provide information concerning the safety after primary administration of live vaccinia virus (LISTER strain). | 1 to 5 years post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (5):
- France (5):
  - Gières
  - Lagord
  - Montpellier
  - Paris
  - Poitiers

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com